CLINICAL TRIAL: NCT00727818
Title: A Split-Blind Clinical Investigation to Compare the Performance and Safety of Inion GTR™ Biodegradable Membrane System to Resorbable Bilayer Bio-Gide®-Membrane of Geistlich Biomaterials in Enhancing Bone Regeneration After Removal of Wisdom Teeth.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Inion Oy (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R304 - 002
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-07

CONDITIONS: Bone Regeneration Following Wisdom Teeth Extraction

INTERVENTIONS:
Device: guided bone regeneration

SUMMARY:
The purpose of this study was to evaluate by histology and histomorphometry, thirty human osseous biopsies sampled from fifteen patients (2 biopsies per patient) following 3 months of implantation. This study is part of a splitting-blind clinical investigation to compare the performance and safety of INION GTRTM Biodegradable Membrane System to resorbable bilayer Bio-Gide®-membrane of Geistlich biomaterials in enhancing bone regeneration after removal of wisdom teeth.

The bone defect and alveolar cavity were augmented with Spongostan® dental 1x1x1cm, Johnson & Johnson, Spreitenbach, Switzerland. The extraction sites were covered on one side with an INION GTRTM Biodegradable Membrane System and on the other with Geistlich resorbable bilayer Bio-Gide®-membrane.

This study was conducted in adaptation to the ISO 10993 Standard : Biological Evaluation of Medical Devices, Part 6 (2007): Tests for Local Effects after Implantation.

This study was conducted in accordance with the requirements of the FDA (Department of health and human services) Good Laboratory Practice (GLP) Regulations, 21 CFR 58 (revised as of April 01, 2005) and in accordance with the requirements of the OECD Good Laboratory Practices, reference ENV/MC/CHEM (98) 17, adapted by council on November 26th 1997.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria: Females or males between the age of 18 to 30 Subject for extraction of both lower fully impacted wisdom teeth Signed informed consent Able and willing to comply with all study procedures

Exclusion criteria: Heavy smoker (>20/day) Insulin dependant diabetes Pregnant or nursing

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-05; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland